CLINICAL TRIAL: NCT06949982
Title: A Randomized Trial To Compare Efficacy And Safety Of Hydroxychloroquine Combined With Methotrexate, Capecitabine And Bevacizumab Versus Regorafenib In Participants With Refractory Metastatic Colorectal Cancer With Mutations In RAS Genes
Brief Title: Efficacy And Safety Of Hydroxychloroquine Combined With Methotrexate, Capecitabine And Bevacizumab Vs. Regorafenib In Participants With Refractory Metastatic Colorectal Cancer With Mutations In RAS Genes
Acronym: x-МАР
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sergey Orlov, MD (Other)
Responsible Party: Sponsor-Investigator, Sergey Orlov, MD, Principal investigator, Pavlov First Saint Petersburg State Medical University
Organization: Pavlov First Saint Petersburg State Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2025-04-14; First posted 2025-04-29 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Colorectal Cancer (mCRC); Colorectal Neoplasms
Keywords: Refractory metastatic colorectal cancer; Hydroxychloroquine; Regorafenib; KRAS mutation; NRAS mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Intervention Model Description: A parallel design is a type of clinical trial in which participants are allocated to two treatment groups: one group receives exclusively one intervention, while the other receives exclusively a different intervention. Randomization in such studies ensures the accuracy of outcomes and reduces the risk of bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group x-MAP (Experimental): This patient cohort will receive systemic therapy with the x-MAP regimen (hydroxychloroquine + methotrexate + capecitabine + bevacizumab) until disease progression or unacceptable toxicity.
  Interventions: Combination Product: experimental group x-MAP
- comparator arm (Active Comparator): This group of patients will receive systemic therapy (regorafenib) according to local standards.
  Interventions: Drug: Regorafenib (BAY 73-4506)

INTERVENTIONS:
Combination Product: experimental group x-MAP — hydroxychloroquine 200 mg TID PO+ methotrexate 2.5 mg BID twice a week PO+ capecitabine 1000 mg/m2 PO BID for 14 days+ bevacizumab 7.5 mg/m2 IV on day 1, every 3 weeks.
  Arms: experimental group x-MAP
Drug: Regorafenib (BAY 73-4506) — Regorafenib 160 mg PO daily on days 1-21, every 28 days OR 1st cycle: Regorafenib 80 mg PO daily on days 1-7, followed by 120 mg PO daily on days 8-14, followed by 160 mg PO daily on days 15-21, every 28 days, 2nd and subsequent cycles: Regorafenib 160 mg PO daily on days 1-21, every 28 days
  Arms: comparator arm

SUMMARY:
This study will evaluate efficacy and safety of hydroxychloroquine combined with methotrexate, capecitabine and bevacizumab versus regorafenib in participants with refractory metastatic colorectal cancer with mutations in KRAS or NRAS genes. The hypotheses of this study are that a combination of hydroxychloroquine, methotrexate, capecitabine, and bevacizumab (compared to regorafenib) prolongs progression-free survival and overall survival, and also increases rates of objective responses and disease control.

DETAILED DESCRIPTION:
One potential therapeutic option for pretreated patients with RAS-positive metastatic colorectal cancer (mCRC) could be hydroxychloroquine. The KRAS mutation drives uncontrolled proliferation and cell survival through pathways such as MAPK/ERK and PI3K/AKT. The pathways in KRAS-mutant tumor cells activate autophagy to recycle cellular components and sustain growth under stress conditions, such as hypoxia or nutrient deprivation. Autophagy serves as a pro-survival mechanism, enabling tumor cells to resist intrinsic stressors and treatment, such as chemotherapy or radiation therapy. Hydroxychloroquine inhibits autophagy by blocking the fusion of autophagosomes with lysosomes. This results in the accumulation of damaged organelles and toxic metabolites within the cell, ultimately triggering apoptosis. Suppressing autophagy may also disrupt tumor cell metabolism by increasing oxidative stress. In experimental models, KRAS-mutant tumors demonstrated enhanced sensitivity to autophagy inhibitors such as hydroxychloroquine. In murine studies, combining hydroxychloroquine with chemotherapy or MAPK pathway inhibitors, such as trametinib, augmented antitumor efficacy. Multiple studies have reported that hydroxychloroquine achieves rapid objective responses when combined with targeted therapy or chemotherapy. However, rapid development of acquired resistance remains a challenge.

Methotrexate and capecitabine may be considered as options for overcoming acquired resistance to hydroxychloroquine. KRAS-mutant tumors frequently exhibit defects in DNA repair systems. Methotrexate inhibits thymidylate synthesis, causing accumulation of DNA damage, especially uracil misincorporation, which leads to "thymidylate-induced stress" and cell death. Cells with mutations in the KRAS gene may have increased expression of folate transporters, such as RFC or FPGS, making them more sensetive to antifolates such as methotrexate. This increases intracellular drug accumulation and cytotoxic effects. Preclinical studies have shown that exposure to methotrexate in tumor cells with KRAS mutations significantly decreases mRNA expression of the KRAS gene and total levels of KRAS protein. When combined with fluoropyrimidines like capecitabine, methotrexate may enhance suppression of DNA synthesis, which is a critical vulnerability in KRAS-mutant tumors.

Capecitabine increases the sensitivity of KRAS-positive tumors to TRAIL-induced apoptosis, a process that may be amplified by hydroxychloroquine exposure. Bevacizumab can be used to improve the delivery of chemotherapy drugs to tumor cells by increasing drug concentration within the tumor through lowering vascular permeability.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Provide written informed consent
* Age ≥ 18 years
* Histologically confirmed diagnosis of colorectal cancer (CRC) with distant metastases.
* Presence of mutations in the KRAS or NRAS gene.
* Participants must have previously treated for metastatic colorectal cancer and experienced disease progression during receiving at least 2 lines of systemic chemotherapy in combination with antiangiogenic agents.
* Patient has previously received oxaliplatin- and irinotecan-containing regimens and developed resistance to these chemotherapeutic agents.

Exclusion Criteria:

* Presence of clinically significant cardiovascular disease: severe or unstable ischemic heart disease, history of myocardial infarction, New York Heart Association Class III/IV congestive heart failure, ventricular arrhythmias.
* Stroke and/or transient ischemic attack within 6 months prior to screening;
* Uncontrolled hypertension
* History of previous malignancies except non-melanoma skin cancers, or in situ cervical or breast cancer unless a complete remission was achieved at least 2 years prior to randomization AND no additional therapy is required during the study period. Patients having hepatic involvement of cancer should be excluded as per investigator assessment.
* Patients with CNS metastases are eligible only if the metastases are adequately treated.
* Absolute neutrophil count (ANC) <1.5×109/L, platelet count <100×109/L, or hemoglobin <9.0 g/dL.
* Serum total bilirubin >1.5 × the upper limit of normal (ULN). Participants with Gilbert syndrome, bilirubin <2 X ULN, and normal AST/ALT are eligible;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × ULN;
* Serum creatinine >1.5 × ULN.
* History of a thromboembolic event
* Presence of any allergic reactions to components of the study drugs
* Concomitant medications with a known risk of causing QT prolongation and/or Torsades de Pointes.
* Any anti-cancer systemic therapy, radiation therapy
* Women who are pregnant or lactating;
* Presence of unresolved adverse events of grade 2 or higher toxicity, according to CTCAE v5.0 criteria, from prior therapy (except for alopecia or neurotoxicity grade≤2).
* Any other serious or uncontrolled medical disorder, active infection, physical examination finding, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a patient's ability to comply with the study requirements, substantially increase risk to the patient, or impact the interpretability of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | From randomization until the first documentation of best overall response (up to 24 months)
  objective response rate (ORR) was defined as the proportion of participants whose best overall outcome included a confirmed complete response (CR) or partial response (PR), assessed by the investigator using RECIST version 1.1 criteria. PR corresponds to a minimum 30% reduction in the total diameter of target lesions compared to the baseline measurements. CR indicates the total disappearance of all identified target lesions. Additionally, any pathological lymph nodes (classified as target or non-target) must shrink to a short axis measurement below 10 millimeters (mm).
Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | From randomization until the first documentation of objective progression or death, whichever comes first (up to 24 months)
  Progression-free survival (PFS) was defined as the time from randomization to the initial occurrence of documented disease progression (PD) or death from any cause, whichever occurs earlier. According to RECIST 1.1 criteria, PD was characterized by at least a 20% enlargement in the total diameter of target lesions compared to the smallest sum recorded during the study, along with an absolute increase of 5 mm or more. The development of any new lesions was also classified as PD.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until the first documentation of objective progression or death, whichever comes first (up to 24 months)
  Overall survival (OS) was measured as the duration (in months) from date of randomization to death resulting from any cause. Participants who had not experienced death by the time of data analysis were censored at their most recent confirmed date of survival.
Disease Control Rate (DCR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | From randomization until the first documentation of objective progression or death, whichever comes first (up to 24 months)
  DCR defined as the proportion of participants with confirmed complete response (CR), partial response (PR), or stable disease (SD) as their best overall response, assessed using RECIST version 1.1 criteria for both target and non-target lesions. PR: A reduction of at least 30% in the total diameter of target lesions relative to the initial baseline measurements. CR: The complete resolution of all identified target lesions. Pathological lymph nodes (target or non-target) must also exhibit a short axis reduction to under 10 mm. SD: Lesions showing neither sufficient shrinkage to meet PR criteria nor sufficient growth to qualify as progressive disease (PD), using the smallest total lesion size recorded during the study as the reference point. PD: Defined as a minimum 20% increase in the total diameter of target lesions compared to the lowest recorded measurement (nadir), which must also include an absolute increase of ≥5 mm. The emergence of new lesions also constitutes PD.
Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | From randomization until the first documentation of objective progression or death, whichever comes first (up to 24 months)
  DOR was measured as the time (in months) from the initial documentation of a partial response (PR) or complete response (CR) according to RECIST version 1.1 criteria until the first confirmed instance of disease progression (PD) or death from any cause, whichever occurred earlier.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs | From start of study drug administration up to approximately 38 months
  An adverse event (AE) refers to any unfavorable or unintended medical event experienced by a participant in a clinical trial involving a medicinal product, regardless of whether it is causally linked to the treatment. A treatment-emergent adverse event (TEAE) was defined as an AE that: began on or after the start of treatment, had an unspecified onset date, existed prior to treatment but worsened in severity after treatment initiation, continuing until 30 days after the final dose of the study drug or the start of subsequent anti-tumor therapy (whichever occurred first). Additionally, serious adverse events (SAEs) deemed treatment-related were classified as TEAEs even if they occurred after this 30-day period. AEs with missing or unreported onset dates were also categorized as TEAEs. Adverse events were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- First Pavlov State Medical University, Saint Petersburg, Sankt-Peterburg, Russia

IPD SHARING:
Plan to Share IPD: No